CLINICAL TRIAL: NCT01178775
Title: Development and Validation of Perceived Fatigue Meaning Scale and Its Effect on Individualized Patient Education and Walking Program for Managing Fatigue in Patients With Cancer
Brief Title: Development and Validation of Perceived Fatigue Meaning Scale on Walking Program
Acronym: PFMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Shiow-Ching Shun/ Assitant Professor, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 200807050R
Record Dates: First submitted 2010-04-11; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Gastric Cancer
Keywords: fatigue; meaning; education; walking program
MeSH Terms: conditions — Stomach Neoplasms; Fatigue | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): control design
- 2 (No Intervention): education only group
- 3 (Experimental): education and education and walking program design
  Interventions: Behavioral: walking

INTERVENTIONS:
Behavioral: walking — use a pedometer for records steps.
  Arms: 3

SUMMARY:
The aims of this three-year study are to:

1. develop and validate a perceived meaning of fatigue scale
2. examine the effect of individualized patient education and walking programs on alleviating fatigue in patients with gastric or colorectal cancer,and further explore the relationship between the perceived meaning of fatigue and intervention outcome.

DETAILED DESCRIPTION:
In the first year, patients will be recruited from oncology inpatient wards and outpatient clinics in two medical center hospitals in Taipei. Purposive sampling will be used to recruit outpatients or inpatients receiving chemotherapy. Data will be analyzed by descriptive analysis, independent t-test, Pearson correlation, one-way analysis of variance, and exploratory factor analysis.

In the second and third years, an experimental design consisting of three groups including a control group, an education only group, and an education and walking program group will be used. Data will be collected at treatment weeks 1, 4,8,12,16 including three cycles of chemotherapy. Data will be analyzed by descriptive analysis, independent t-test, Pearson correlation, and generalized estimating equations. At least 230 subjects will be interviewed in the first year.

At least 105 of patients with gastric cancer or colorectal will be classified into the three groups in the second and third year. We expect the results of this study to explore the meaning of fatigue and to help develop a common strategy to manage fatigue in Taiwan. The results can help clinicians and researchers to tailor interventions for cancer patients with severe fatigue.

ELIGIBILITY:
Inclusion Criteria:

* The patients with gastric cancer during receiving chemotherapy
* Those who are willing to participate in the research
* Aged above 18

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue Symptom Inventory | Time point(s) at which outcome measure is assessed at 16 Weeks after recruting in this study .
  the level of fatigue in three groups will be measured at the end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, Ph.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan